CLINICAL TRIAL: NCT07231406
Title: A Cluster Randomized Controlled Trial of Narrative Therapy Among Young People With Moderate Level of Mental Distress in Hong Kong
Brief Title: Narrative Therapy Among Young People With Moderate Level of Mental Distress in Hong Kong
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); The Boys' and Girls' Clubs Association of Hong Kong (Other); Caritas Medical Centre, Hong Kong (Other); Hong Kong Christian Service (Other); Neighbourhood Advice-Action Council (Other); St. James' Settlement (Other); Tung Wah Group of Hospitals (Other); Hong Kong Young Women's Christian Association (Other); Yan Oi Tong (Unknown); The Salvation Army, Hong Kong and Macau Command (Other); Hong Kong Playground Association (HKPA) (Unknown); Hong Kong Sheng Kung Hui Welfare Council Limited (Other); Hong Kong Children and Youth Services (HKCYS) (Unknown); Hong Kong Federation of Youth's Group (HKFYG) (Other); Chinese YMCA of Hong Kong (Unknown)
Responsible Party: Principal Investigator, Dr. Christy Lai-ming Hui, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250818-006-000
Record Dates: First submitted 2025-08-27; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Mental Distress
Keywords: cluster randomized controlled trial; narrative therapy; youths; mental distress
MeSH Terms: interventions — Narrative Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NT Intervention (Active Comparator): This narrative therapy intervention will: (i) facilitate shared experiences among participants, (ii) support the reconstruction of personal identity, (iii) promote collective wisdom-sharing and skill development; and (iv) foster solidarity in imagining diverse life possibilities. This approach empowers young people to critically engage with dominant narratives and discover their own authentic paths. The NT intervention consists of six sessions, conducted in a small-group format (6 - 8 participants per group). Youths at similar life stages, such as secondary students, university students, and early-career young professionals, will be grouped together to encourage meaningful discussions and shared experiences. The program consists of six sessions, with the first five lasting 1.5 hours each, and the final session (Section 6) extending to 2 hours for a comprehensive closing. All sessions will be conducted face-to-face by frontline social or youth workers who have received prior training,
  Interventions: Behavioral: Narrative Therapy
- Waitlist Control (No Intervention): Participants allocated to the waitlist control group will wait for 10 weeks (6 + 4 weeks) before receiving the NT intervention

INTERVENTIONS:
Behavioral: Narrative Therapy — In Hong Kong, deeply ingrained norms and expectations shape each stage of life. As young people navigate their growth, they are constantly influenced by mainstream narratives stemming from sociocultural traditions, family, educators, peers, or social media. These narratives often define socially approved notions of "good" versus "bad," "meaningful" versus "meaningless," and "successful" versus "failing." Many youths may not fully realize how these dominant discourses subtly influence their life choices, often leading them to unconsciously accept predetermined paths they believe they "should" follow. Whether they conform successfully or struggle with these expectations, young people frequently experience pressure and negative emotions. Even more concerning, some internalize these societal judgments, resulting in negative self-perceptions. Through this group program utilizing narrative intervention methods, we aim to provide a safe, supportive space for youth to re-examine and explore th
  Arms: NT Intervention

SUMMARY:
This cluster randomized controlled trial (cRCT) aims to evaluate the effectiveness of a narrative therapy (NT) intervention in (i) reducing mental distress, depressive symptoms, and anxiety, as well as (ii) enhancing perceived control and fostering a stronger sense of self among at-risk youth in Hong Kong. Participants are youths with moderate mental health concerns, indicated by K6 scores ranging from 11 to 14.

The study involves seven clusters, each based on community hubs, which will be randomly assigned to either the intervention group or a wait-list control group. Clusters assigned to the intervention group will receive six face-to-face sessions led by trained youth workers. Control clusters will receive the same intervention after the initial follow-up period.

Participants will be evaluated at baseline, post-intervention, and one-month follow-up. An interim analysis is built for the sake of evaluation of the collected data from the ongoing trial, in which the primary research question is addressed, and which has the potential for modifying the conduct of the study. Furthermore, a qualitative follow-up will be conducted after the trial, involving both participants and the workers delivering the NT intervention. This qualitative component aims to gather feedback on participants' experiences, and inform potential revisions to enhance future implementation.

It is hypothesized that youths receiving the NT intervention will show significantly greater improvements in perceived control and sense of self, along with reductions in mental distress, as well as depressive and anxiety symptoms, compared to those in the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* JC LevelMind @ Community users at risk for mental distress (Tier 2), with K6 scores ranging from 11 to 14
* Aged between 12 and 24 years
* Sufficiently proficient in Chinese to comprehend verbal instructions
* Able to provide written informed consent (parental consent for participant aged 12-17)

Exclusion Criteria:

* Known diagnosis of intellectual disability
* Organic brain disorder
* Established psychiatric diagnosis
* Current substance abuse
* Receiving other structured psychological therapies such as module-based psychological therapy, mentalization-based therapy, low-intensity online interventions, cognitive-behavioral therapy, cognitive-behavioral therapy for insomnia, mindfulness, or art-informed therapy within the hub setting or any others outside the hub setting
* Presence of current or active suicidal ideation or attempts

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 770 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | Baseline, 6-week, and 10-week
  The 6-item Kessler Psychological Distress Scale (scores range from 0 to 24 where a higher score indicates a worse outcome)
Depression and anxiety Symptoms | Baseline, 6-week, and 10-week
  Depression Anxiety Stress Scales (scores range from 0 to 63 where a higher score indicates more severe symptoms)
Perceived Control / Self-efficacy | Baseline, 6-week, and 10-week
  Sense of Mastery Scale (scores range from 7 to 28 where a higher score indicates a a better outcome)

SECONDARY OUTCOMES:
Narrative Identity | Baseline, 6-week, and 10-week
  Narrative Identity Self-Evaluation Scale (scores range from 0 to 200 where a higher score indicates a better outcome)
Perceived Social Support | Baseline, 6-week, and 10-week
  Multidimensional Scale of Perceived Social Support (scores range from 12 to 84 where a higher score indicates a better outcome)
Loneliness | Baseline, 6-week, and 10-week
  UCLA Loneliness Scale (scores range from 20 to 80 where a higher score indicates a worse outcome)
Resilience | Baseline, 6-week, and 10-week
  The 10-item Connor-Davidson Resilience Scale (scores range from 0 to 40 where a higher score indicates a better outcome)
Rumination | Baseline, 6-week, and 10-week
  The 22-item Rumination-Reflection Questionnaire (scores range from 22 to 88 where a higher score greater rumination)
Self-stigma | Baseline, 6-week, and 10-week
  The 9-item Internalized Stigma of Mental Illness Inventory (scores range from 1 to 4 where a higher score indicating high internalized stigma)
Hopefulness / Hopelessness | Baseline, 6-week, and 10-week
  Beck Hopelessness Scale (scores range from 0 to 20 where a higher score indicates greater levels of hopelessness)
Service Utilization | Baseline, 6-week, and 10-week
  Client Service Receipt Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Christy Lai Ming Hui, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No